CLINICAL TRIAL: NCT00326157
Title: Phase II Pilot Study on Safety of Administration of 3mg/kg/Day Three Times a Week Until Day 22 (21 Days After Transplantation Day) and 7 mg/kg Weekly From Day 29 to the End of Treatment (Day 50-8th Week) of AmBisome® in Antifungal Primary Prophylaxis Treatment of High Risk Patients Undergoing Allogeneic Stem-cell Transplantation
Brief Title: PROPHESSOR: AmBisome in Antifungal Primary Prophylaxis Treatment of High Risk Patients Undergoing Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Luigi Antonio Picaro, Gilead Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS-IT-131-0151
Record Dates: First submitted 2006-05-10; First posted 2006-05-16 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Fungus Diseases
Keywords: antifungal primary prophylaxis treatment; allogeneic stem-cell transplantation; antifungal primary prophylaxis treatment of high risk patients undergoing allogeneic stem-cell transplantation
MeSH Terms: conditions — Mycoses | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AmBisome® will be administered for a duration of 8 weeks
  Interventions: Drug: AmBisome

INTERVENTIONS:
Drug: AmBisome — 3mg/kg/day three times a week until day 22 (21 days after transplantation day) and 7 mg/kg weekly from day 29 to the end of treatment (day 50-8th Week) of AmBisome®, IV administration

SUMMARY:
This pilot study was designed in order to evaluate the safety and efficacy of an AmBisome® loading dose regimen, in a weekly administration schedule during the initial phase of allogeneic stem-cell transplant and in case of occurrence of graft versus host disease (GvHD), which are both high risk periods as far as severe fungal infection development is concerned.

DETAILED DESCRIPTION:
This pilot study was designed in order to evaluate the safety and efficacy of an AmBisome® loading dose regimen, in a weekly administration schedule during the initial phase of allogeneic stem-cell transplant and in case of occurrence of GvHD, which are both high risk periods as far as severe fungal infection development is concerned.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged more than 18 years
* Patients with hematological malignancies undergoing allogeneic stem cell transplantation from donors other than human leukocyte antigen (HLA) identical sibling; source of stem cell includes either peripheral blood or bone marrow
* No evidence of fungal infection at chest computed tomography (CT) scan and at sinus X-ray at baseline
* Patients with no sign or symptoms of fungal infection and no previous proven or probable invasive fungal infection (IFI)
* Females of childbearing potential must be surgically incapable of pregnancy, or practising a method of birth control, or agree to abstain from heterosexual intercourse while participating in the study, and with a negative pregnancy test (blood or urine) at baseline
* An understanding of the study and agreement of the patient to give written informed consent
* Ability and agreement to comply with all study requirements
* Patient willing to attend hospital appointments for each injection (infusions will be performed in the hospital, under strict medical supervision). All patients will be hospitalised prior to, and remain in the hospital for at least one day, after the first infusion.

Exclusion Criteria:

* Known hypersensitivity to amphotericin B, in particular known history of anaphylactic reaction to amphotericin B
* Patients undergoing cord transplantation
* Creatinine > 2.0 mg/dL
* Patient with moderate or severe liver disease as defined by AST or ALT > 5 times the upper limit of normal (ULN)
* Patients who are unlikely to survive more than 1 month
* Patients who have received systemic antifungal therapy within 15 days prior to the inclusion
* Any severe cardiovascular disease (such as arrhythmias, in particular) which may constitute a contra-indication to AmBisome® administration
* Any severe disease other than the hematological diseases described at the second point of inclusion criteria, which in the investigator's judgement may interfere with study evaluations or affect the patient's safety
* Pregnant or nursing females
* Patients previously included in this study
* Patients who have taken any investigational drug in the last 30 days prior to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile will be obtained by considering: Number (%) of patients with adverse events (AEs) | Through 16 weeks
Number (%) of patients with infusion related AE | Through 16 weeks
Laboratory parameters (in particular renal toxicity, hepatotoxicity, hypokalaemia, hypomagnesaemia) | Through 16 weeks
Overall adverse events | Through 16 weeks

SECONDARY OUTCOMES:
Number (%) of patients with probable or proven invasive fungal infection according to EORTC-MSG criteria within the 6 months following the initiation of prophylaxis treatment | Within previous 6 months
Number (%) of patients with fever of unknown origin requiring empirical antifungal treatment within the 6 months following the initiation of prophylaxis treatment | Within previous 6 months
Number (%) of patients with superficial fungal infections within the 6 months following the initiation of prophylaxis treatment | Within previous 6 months
Number (%) of patients with evidence of colonization by fungal organisms observed within the 6 months following the initiation of prophylaxis treatment | Within previous 6 months
Reasons for early study discontinuation | Through 16 weeks
Survival rate and incidence of mortality related to fungal infection at the end of treatment and within 3, 6, and 12 months after the initiation of prophylaxis treatment | Within 12 months
Time to probable or proven invasive fungal infection; fever of unknown origin requiring empirical antifungal treatment | Through 16 weeks
Time to superficial fungal infections | Through 16 weeks
Time to initiation of empirical antifungal treatment | Through 16 weeks
Time to study discontinuation | Through 16 weeks
Number of patients enrolled | Through 16 weeks
Number of patients completing the study | Through 16 weeks
Number of patients with early discontinuation | Through 16 weeks
Number of patients classified by reason for discontinuing study drug (including the study completion) | Through 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Picaro, MD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Milan, Italy